CLINICAL TRIAL: NCT00003514
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Metastatic or Incurable Neuroendocrine Tumors
Brief Title: Antineoplaston Therapy in Treating Patients With Neuroendocrine Tumor That Is Metastatic or Unlikely to Respond to Surgery or Radiation Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-NE-2; CDR0000066557 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Merkel Cell Carcinoma; Islet Cell Carcinoma; Neuroendocrine Carcinoma; Pituitary Tumor
Keywords: ACTH-producing pituitary tumor; prolactin-producing pituitary tumor; growth hormone-producing pituitary tumor; recurrent pituitary tumor; TSH producing pituitary tumor; nonfunctioning pituitary tumor; somatostatinoma; stage III Merkel cell carcinoma; recurrent Merkel cell carcinoma; neuroendocrine carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell; Carcinoma, Islet Cell; Carcinoma, Neuroendocrine; Pituitary Neoplasms; Growth Hormone-Secreting Pituitary Adenoma; Somatostatinoma | interventions — antineoplaston A10; antineoplaston AS 2-1; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally-occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating patients with neuroendocrine tumor that is metastatic or unlikely to respond to surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide treatment with antineoplastons A10 and AS2-1 for patients with metastatic or incurable neuroendocrine tumors.
* Describe response, tolerance to, and side effects of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gradually escalating doses of antineoplastons A10 and AS2-1 by intravenous injection 6 times daily until the maximum tolerated dose is reached.

Treatment continues for at least 2 months in the absence of unacceptable toxicity or disease progression. Patients achieving complete response (CR) continue treatment for an additional 8 months after reaching CR.

Tumors are measured every 2 months for 1 year and then every 3 months for 1 year.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable neuroendocrine tumor that is unlikely to respond to existing therapy, meeting 1 of the following criteria:
* Metastatic disease
* Disease that is not curable with surgery or radiotherapy
* Measurable disease by MRI or CT scan
* Tumor must be at least 2 cm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* No renal insufficiency
* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection
* No concurrent nonmalignant systemic disease
* Not a high medical or psychiatric risk

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy

Surgery:

* Recovered from prior surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplastons
* No other concurrent antineoplastic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States